CLINICAL TRIAL: NCT07235800
Title: The Effect of Virtual Reality-Based Episiotomy Simulation on Midwifery Students' Skills and Self-Efficacy Levels
Brief Title: VR Episiotomy Simulation: Impact on Midwifery Students' Skills and Self-Efficacy (VESES)
Acronym: VESES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Collaborators: Inonu University (Other)
Responsible Party: Principal Investigator, Sibel Akgül Kartal, Lecturer, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025/17627; TDK-2020-2165 (Other Grant/Funding Number: Inonu University Scientific Research Projects Coordination Unit (BAP))
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Use of Virtual Reality Simulation in Midwifery Training
Keywords: Midwifery Virtual Reality Simulation Episiotomy Learning Process

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the virtual reality simulation group or the traditional mannequin training group. Both groups receive the same theoretical education, followed by their respective practical training interventions in parallel.
Who Masked: Participant
Masking Description: No blinding (masking) was applied in this study. Participants were unaware of their group allocation only during the initial training session, but by the time of the one-month follow-up data collection, they were aware of their group assignment. Instructors and outcome assessors were aware of group assignments throughout the study."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Simulation Group (Experimental): Participants in this group will receive episiotomy skills training using a virtual reality (VR) simulation environment. The training will include a theoretical session followed by hands-on practice in a simulated virtual birth room using VR equipment.
  Interventions: Behavioral: Virtual Reality Simulation Training
- Control Group (Active Comparator): Participants in this group will receive episiotomy skills training using traditional silicone-based episiotomy mannequins. The training includes the same theoretical content as the intervention group, followed by hands-on practice using anatomical models.
  Interventions: Behavioral: Traditional Episiotomy Training

INTERVENTIONS:
Behavioral: Virtual Reality Simulation Training — This intervention is a virtual reality (VR)-based episiotomy simulation designed for midwifery students. The training is conducted in an immersive virtual delivery room, where participants perform the steps of episiotomy incision and suturing using VR headsets, motion sensors, and hand controllers. The simulation includes virtual surgical tools and interactive elements that replicate a clinical environment. This VR-based training differs from traditional model-based education by providing a more engaging and realistic experience, aiming to improve students' psychomotor skills and self-efficacy in performing episiotomy.
  Other Names: VR Episiotomy Simulation; Virtual Reality-Based Episiotomy Training; VR Episiotomy Skills Training
  Arms: VR Simulation Group
Behavioral: Traditional Episiotomy Training — This intervention consists of a traditional episiotomy training session using physical anatomical models (manikins) in a classroom environment. The training includes hands-on practice of episiotomy incision and suturing on silicone-based or synthetic perineal models, supervised by the instructor. This method reflects standard educational practices in midwifery training and does not involve virtual reality or simulation technology.
  Other Names: Conventional Episiotomy Education; Episiotomy Model Training
  Arms: Control Group

SUMMARY:
This study aims to develop and evaluate a virtual reality (VR)-based episiotomy training simulation for midwifery students. Episiotomy is a surgical procedure performed during childbirth, and incorrect application may lead to serious psychological and physiological consequences. While traditional training methods often use animal tissues or synthetic materials, recent advances in technology have introduced simulation-based learning. VR technology has shown potential to enhance learning outcomes, confidence, and satisfaction among healthcare students. Despite its growing use in medical education, there is currently no VR training model specifically designed for teaching episiotomy skills. This study will design a VR episiotomy simulation, assess its effectiveness in skill acquisition and learning, and propose it as a new educational method in midwifery training.

DETAILED DESCRIPTION:
This study aims to develop and evaluate a virtual reality (VR)-supported episiotomy simulation training program for midwifery students. The unique contribution of this study lies in assessing skills acquisition, learning processes, and satisfaction differences in VR-based episiotomy training, a field where no previous VR applications for episiotomy skills training have been identified in the literature.

A randomized controlled parallel-group design will be employed. The study will take place at Van Yuzuncu Yıl University Faculty of Health Sciences (YYU FHS) between April 2025 and April 2026. The episiotomy topic is covered theoretically and practically within the Risky Birth and Postpartum Course for third-year midwifery students at YYU FHS. Currently, mannequin models are used for episiotomy practice.

The study population will consist of third-year midwifery students at YYU FHS, totaling 90 students. The sample will be composed of students who voluntarily agree to participate and meet inclusion criteria. Sample size was calculated using G*Power 3.1.9.2 software based on the primary dependent variable-mean self-efficacy scores-yielding a minimum of 38 students per group (VR intervention and control groups), with an effect size of 0.50, power of 0.95, and alpha of 0.05. Participants will be randomized equally into two groups using the Random.org platform to prevent selection bias.

Inclusion criteria are: proficiency in Turkish, no prior episiotomy training, and no medical contraindications for VR use (e.g., epilepsy).

Data collection tools include:

Demographic Information Form

Skill Evaluation Form

Episiotomy Skills Self-Efficacy Scale (EBÖÖ)

Student Satisfaction Survey

Data collection will be performed by an independent researcher who is not involved in the intervention delivery or study design. Due to the visible nature of the intervention (VR headset vs. mannequin), full blinding of the outcome assessor is not feasible. However, all evaluations will be conducted using standardized assessment tools to reduce observer bias and ensure objectivity. Assessments will occur pre-training, immediately post-training, and one month after training.

The intervention includes a two-day training program. On the first day, all students receive four hours of theoretical instruction on episiotomy. On the second day, the control group practices on traditional mannequins for four hours, while the intervention group trains using the VR simulation for the same duration. The VR simulation immerses students in a virtual delivery room where they perform episiotomy and repair using virtual surgical tools and equipment.

The VR setup includes VR goggles, two control handles, motion sensors, and a high-performance computer. The episiotomy mannequin used in the control group realistically simulates perineal anatomy for skill practice.

Dependent variables are students' skill performance and self-efficacy scores; the independent variable is the VR-supported episiotomy training.

Study limitations include the single-center design with only YYU third-year students and the high cost of VR software and equipment.

Data will be analyzed using SPSS 25. Descriptive statistics (mean, standard deviation) and inferential tests (independent and paired sample t-tests) will be conducted to evaluate group differences and within-group changes.

This study is expected to demonstrate the feasibility and effectiveness of VR technology in enhancing midwifery education and propose an innovative training tool for episiotomy skills development.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and understand Turkish

Have not received previous episiotomy training

No medical conditions preventing the use of virtual reality (e.g., epilepsy)

Enrolled as a third-year midwifery student at Van Yüzüncü Yıl University Faculty of Health Sciences

Exclusion Criteria:

* Individuals who do not speak or understand Turkish

Those who have previously received episiotomy training

Participants with medical conditions contraindicating the use of virtual reality (e.g., epilepsy)

Not enrolled as a third-year midwifery student at Van Yüzüncü Yıl University Faculty of Health Sciences

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2025-12-21 (Estimated); Primary Completion 2026-01-22 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Episiotomy Self-Efficacy Score | Baseline (before training), immediately after training, and 1 month after training
  Participants' episiotomy-related self-efficacy will be assessed using the Episiotomy Skills Self-Efficacy Scale (EBÖÖ), a validated 19-item Likert-type instrument. Each item is scored from 1 (strongly disagree) to 4 (strongly agree), with total scores ranging from 19 to 76. Higher scores indicate greater self-efficacy.

SECONDARY OUTCOMES:
Episiotomy Skill Performance Score | Immediately after training
  Participants' practical episiotomy skills will be evaluated through a researcher-developed checklist. This checklist covers key steps in the episiotomy procedure. Each step is observed and scored, providing a total
Student Satisfaction with Training Method | Immediately after training and 1 month after training
  Participants' satisfaction with the training method (VR or traditional mannequin) will be assessed using a researcher-developed satisfaction questionnaire. This includes Likert-scale questions evaluating the perceived usefulness, engagement, and satisfaction with the training.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel AKGÜL KARTAL, Lecturer, Principal Investigator — Yuzuncu Yil University, Faculty of Health Sciences
Locations (1):
- Van Yüzüncü Yıl University Faculty of Health Sciences, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The plan to share individual participant data is still under consideration and will depend on institutional policies and participant consent.

REFERENCES:
- See also: Related Info — https://tez.yok.gov.tr/UlusalTezMerkezi/tezDetay.jsp?id=63801